CLINICAL TRIAL: NCT00126789
Title: An Open-Label, Long-Term Safety Study to Evaluate the Safety of the ZR-02-01 Matrix Transdermal Fentanyl Patch for the Treatment of Moderate to Severe Cancer Pain
Brief Title: Fentanyl Transdermal Matrix Patch ZR-02-01 to Treat Moderate to Severe Cancer Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Based on PK data, product did not meet requirement for further development.
Sponsor: ZARS Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZMF-301
Record Dates: First submitted 2005-08-02; First posted 2005-08-04 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Pain; Cancer
Keywords: Pain Cancer; Chronic Pain
MeSH Terms: conditions — Pain; Neoplasms; Cancer Pain; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ZR-02-01 (Experimental): ZR-02-01 matrix transdermal fentanyl patch
  Interventions: Drug: Fentanyl Transdermal Matrix Patch ZR-02-01

INTERVENTIONS:
Drug: Fentanyl Transdermal Matrix Patch ZR-02-01 — ZR-02-01 patch contains fentanyl dispersed in a solid matrix, and will be available in 25, 50, 75 and 100 mcg/hr patches. The patches will be worn on the chest or upper arm and an overlay will be placed over the patch. Patches (and overlays) will be replaced every 3 days by the patient and/or responsible caregiver. If a patient experiences end-of-dose-failure, the dosing interval may be changed by the physician investigator to every 2 days. The maximum dose allowed in this study is 300 mcg/hr.
  Other Names: ZR-02-01 matrix transdermal fentanyl patch

SUMMARY:
The purpose of this study is to evaluate the safety of the matrix fentanyl patch ZR-02-01 in providing relief of cancer pain.

DETAILED DESCRIPTION:
This study will evaluate the safety of the matrix fentanyl patch. The study will be conducted in opioid-tolerant patients with moderate to severe cancer pain currently taking an around-the-clock opioid. Patients will discontinue their current opioid regimen and begin using ZR-02-01 as soon as possible under the direction of the physician investigator upon entry into the study. Patient's dose of ZR-02-01 will be determined by the investigator using sponsor-provided conversion. Pain therapy will be under the supervision of the physician investigator.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 and no older than 75 years of age at the time of screening
* Patient has a diagnosis of cancer
* Patient has moderate to severe pain that is related to cancer or its treatment and is expected to last indefinitely and is currently taking an around-the-clock opioid to treat his/her pain
* Patient is already receiving opioid therapy, has demonstrated opioid tolerance
* A responsible adult caregiver is available in the event of an emergency at home

Exclusion Criteria:

* Patient has uncontrolled or rapidly escalating pain as determined by the investigator
* Patient has a history of substance abuse or has a substance abuse disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-08; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 12 weeks
  To evaluate the safety of long-term administration of the ZR-02-01 patch for the treatment of moderate to severe cancer pain

SECONDARY OUTCOMES:
Pain intensity | 12 weeks
  Patient's evaluation of pain intensity using the VAS (100 mm)
Global Satisfaction satisfied) | 12 weeks
  Global Satisfaction using a 5-point Likert scale (0= not satisfied to 4 = completely satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Rauck, MD, Principal Investigator — The Center for Clinical Research
Locations (2):
- United States (2):
  - Loma Linda Center for Pain Management, Loma Linda, California
  - The Center for Clinical Research, Winston-Salem, North Carolina